CLINICAL TRIAL: NCT06410976
Title: Prospective Clinical Assessment Study in Children With Hypochondroplasia: ACCEL
Brief Title: Prospective Clinical Assessment Study in Children With Hypochondroplasia
Acronym: HCH
Status: Recruiting | Type: Observational
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Other Study IDs: QBGJ398-004
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Hypochondroplasia
Keywords: skeletal dysplasia; endochondral ossification; hypochondroplasia; HCH; shortened proximal limbs; fibroblast growth factor receptor 3; FGFR3; endochondral bone formation; disproportionate short stature; quality of life; dwarfism; bone diseases; musculoskeletal diseases; osteochondrodysplasia; functional abilities; annualized growth velocity; annualized height velocity; growth; genetic diseases; congenital; AHV; AGV
MeSH Terms: conditions — Hypochondroplasia; Mucopolysaccharidosis IV; Dwarfism; Bone Diseases; Musculoskeletal Diseases; Osteochondrodysplasias; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Collect blood for central assessment of blood biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a long-term, multicenter, non-interventional study of children ages 2.5 to <17 years with hypochondroplasia (HCH).

DETAILED DESCRIPTION:
The objective is to evaluate growth, HCH-related medical complications, health-related quality of life, functional abilities and cognitive functions of study participants. Data collected will contribute to the characterization of the natural history of children with HCH. No study medication will be administered.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent.

Aged 2.5 to <17 years at study entry.

Diagnosis of HCH documented clinically by the presence of disproportionate short stature and confirmed with a molecular test.

Participants are ambulatory and able to stand without assistance.

Study participants and parent(s), guardian(s), or caregiver(s) are willing and able to comply with study visits and study procedures.

Exclusion Criteria:

Have ACH or short stature condition other than HCH.

In females, having had their menarche. Annualized height growth velocity ≤1.5 cm/year over a period ≥6 months prior to screening.

Having a clinically significant disease or condition that in view of the investigator or Sponsor will interfere with the evaluation of growth, with study participation or not be in the best interest of the participant.

Clinically significant abnormality in any laboratory test result at screening

Current evidence of corneal or retinal disorders.

Have used any other investigational or approved product or medical device for the treatment of HCH or short stature for ≥ 30 days or with the last dose <6 months before screening.

Have had regular long-term treatment (>1 month) with oral corticosteroids (low-dose ongoing inhaled steroid for asthma is acceptable).

Previous limb-lengthening surgery or guided growth surgery with plates still in place or removed within the 6 months prior to screening.

Having had a fracture of the long bones or spine within 12 months of screening.

History and/or current evidence of extensive ectopic tissue calcification.

History of malignancy.

Concurrent circumstance, disease, or condition that, in the view of the investigator and/or sponsor, would interfere with study participation, and/or would place the participant at high risk for poor compliance with study activities or for not completing the study.

Current participation in any other ongoing clinical study with another sponsor.

Ages: 30 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with hypochondroplasia
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Annualized height velocity | up to 3 years

SECONDARY OUTCOMES:
Change over time in height Z-score, upper arm to forearm ratio, and upper leg to lower leg ratio | up to 3 years
Cognitive functions | up to 3 years
HCH-related medical events reported as medical history or NT-AEs | up to 3 years
HCH-related surgical procedures | up to 3 years
Change from BL in the Physical Functioning dimension of the Pediatric Quality of Life Generic Core Scale Short Form. | up to 3 years
  Scale scores 0-100. Higher score=better Health-Related Quality of Llife

OTHER OUTCOMES:
Change from BL in collagen X marker concentration (ug/L). | up to 3 years

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Madison - Waisman Center Bone Dysplasia Clinic, Madison, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Canada (3):
  - London Health Sciences Centre - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario
  - Université de Montréal - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (3):
  - Hôpital Femme Mère Enfant HCL, Bron
  - Hôpital Necker-Enfants Malades, Paris
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hôpital des Enfants, Toulouse
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Paediatric Clinical Research Unit at Oslo University Hospital, Oslo
- Hospital Pediátrico de Coimbra, Coimbra, Portugal
- KK Women's and Children's Hospital, Singapore, Singapore
- Hospital Vithas San Jose, Vitoria-Gasteiz, Spain
- Astrid Lindgren Children's Hospital, Solna, Sweden
- United Kingdom (4):
  - The Portland Hospital for Women and Children, London, England
  - Manchester University, Manchester, England
  - Sheffield Children's NHS Foundation Trust, Sheffield, England
  - Glasgow Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No